CLINICAL TRIAL: NCT04114383
Title: Concurrent Assessment of Skeletal Muscle Mass and Synthesis/Breakdown in Old Age: Defining Diagnostics and the Aetiology of Sarcopenia to Identify "At-risk" Individuals and Appropriate Countermeasures
Brief Title: Concurrent Assessment of Skeletal Muscle Mass and Synthesis/Breakdown in Old Age
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Abbeyfield (Unknown)
Responsible Party: Sponsor
Other Study IDs: Abbeyfield
Record Dates: First submitted 2019-02-05; First posted 2019-10-03 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-10

CONDITIONS: Sarcopenia; Muscle Atrophy
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy | interventions — Deuterium Oxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: D3-Creatine — 30mg D3-Creatine to measure muscle mass
Other: Deuterium Oxide — D2O provided to measure muscle protein synthesis
  Other Names: D2O; Heavy water
Other: D3-3-methylhistidine — D3-3-methylhistidine is provided to measure muscle protein breakdown
  Other Names: D3-3MH

SUMMARY:
This study involves minimally-invasive techniques to measure muscle mass, muscle protein breakdown and synthesis simultaneously in older age.

DETAILED DESCRIPTION:
Most people will have noticed that with age people become frail. This is principally due to wasting of skeletal muscle known as "sarcopenia". Crucially, sarcopenia is more than just a symptom of weakness and poor functional capacity; it exposes people to an increased risk of falls and fractures, impacting quality of life, independence, health status and ultimately lifespan. Muscles represent the largest organ in the body, making up over 50% of total body weight. Most people know that skeletal muscles are important for movement and to support the skeleton, but not everyone is aware of how important muscles are for whole-body health. For example, muscles represent a vast protein store containing amino acids (the building blocks of protein) which can be broken down in times of fasting, infection and disease in order to provide energy to help other vital organs. Because of the detrimental effects on health, and the associated health costs, sarcopenia is of grave concern. Therefore, there is a significant clinical need to pre-identify at-risk older individuals who have low muscle mass so that they can be offered an intervention (of diet, exercise or drug-based) before they suffer any of the potential problems outlined above. Current techniques for measuring whole-body muscle mass, including MRI and CT are time-consuming, expensive and in huge demand in hospital settings, meaning that muscle wasting conditions such as sarcopenia often go undiagnosed. In this project we propose a potential solution to this problem by developing a diagnostic of sarcopenia that requires only a single drink and subsequent urine collection. In addition, throughout this project we aim to explore the mechanisms underlying muscle wasting by assessing the muscle of those with low and 'normal' muscle mass.

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteers of normal body mass index (BMI <35 kg/m2), aged 65-85 years

Exclusion Criteria:

* A BMI > 35 kg/m2
* Active cardiovascular disease:

  o angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt, recent cardiac event
* Cerebrovascular disease:

  o previous stroke, aneurysm (large vessel or intracranial), epilepsy
* Respiratory disease including:

  o pulmonary hypertension, COPD
* Metabolic disease:

  o hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, type 1 or 2 diabetes
* Active inflammatory bowel or renal disease
* Malignancy
* Recent steroid treatment (within 6 months) or hormone replacement therapy
* Clotting dysfunction

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Generally healthy older adults
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Measurement of D3-Creatine in Urine: 24 hours | Up to 24 hours
  To use 30mg of D3-Creatine to measure muscle creatine pool size (g) and whole-body muscle mass (kg) from urine samples taken between 0 and 72 hours. The 0-24 hours collection provides a measure of creatine spillover.
Measurement of muscle mass using D3-Creatine: 48 hours | 48 hours
  To use 30mg of D3-Creatine to measure muscle creatine pool size (g) and whole-body muscle mass (kg) from urine samples taken between 0 and 72 hours. The 0-24 hours collection provides a measure of creatine spillover, spot urines at 48 and 72 hours provide a measurement of the dilution of tracer in urinary creatinine and thus the total muscle creatine pool size.
Measurement of muscle mass using D3-Creatine: 72 hours | 72 hours
  To use 30mg of D3-Creatine to measure muscle creatine pool size (g) and whole-body muscle mass (kg) from urine samples taken between 0 and 72 hours. The 0-24 hours collection provides a measure of creatine spillover, spot urines at 48 and 72 hours provide a measurement of the dilution of tracer in urinary creatinine and thus the total muscle creatine pool size.
Rate of dilution of D3-3MH by endogenous unlabelled 3MH release in blood | 6 hours (from 24 through to 30 hours)
  Using 10mg of D3-3-methylhistidine (D3-3MH) and subsequent multiple blood sampling between 24 and 30h, the rate of dilution of D3-3MH by endogenous unlabelled 3MH release provides a measure of the rate of whole-body muscle protein breakdown.
Rates of Muscle Protein Synthesis | 3 days
  Using D2O, rate of muscle protein synthesis will be calculated, cumulatively, over 0-3 days by measuring deuterium labelling of alanine into protein from a muscle biopsy at 72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Derby Hospital Medical School, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided